CLINICAL TRIAL: NCT03414060
Title: Feasibility of the Menstrual Cup for Non-Surgical Management of VVF Among Women Seeking Care at a Health Facility in Ghana
Brief Title: Feasibility of the Menstrual Cup for VVF
Acronym: FMCVVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ghana Medical School (Other)
Collaborators: New York University College of Global Public Health (Unknown); NYU Langone Health (Other); Korle-Bu Teaching Hospital, Accra, Ghana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHS-Et/M.9-P3.2/2015-2016
Record Dates: First submitted 2018-01-19; First posted 2018-01-29 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Vaginal Fistula; Vesico Vaginal Fistula; Obstetric; Injury
Keywords: obstetric fistula; vesicovaginal fistula; menstrual cup; pad test; non-surgical management; feasibility; acceptability; innovation; coping; incontinence
MeSH Terms: conditions — Vaginal Fistula; Vesicovaginal Fistula; Wounds and Injuries | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Intervention Model Description: repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Menstrual Cup) (Experimental): The menstrual cup is a 100% silicone, flexible reservoir cup that, when inserted correctly in the vagina, is sanitary and efficacious in preventing leakage of menstrual blood and in eliminating odor.
  Interventions: Device: Menstrual Cup

INTERVENTIONS:
Device: Menstrual Cup

SUMMARY:
This study examines the feasibility and acceptability of the vaginal menstrual cup for short-term management of vesicovaginal fistula (VVF) among 11 women seeking treatment at a health facility in Ghana. The repeated measures design utilizes a 2-hr pad test to compare urinary leakage with and without the insertable cup, a questionnaire on acceptability and perceived effect is administered and a clinical exam is completed. Subsequently, semi-structured interviews will be carried out with up to 24 additional women seeking treatment at a health facility in Ghana. Interviews will cover women's experiences of living with fistula, including strategies for coping with urinary incontinence and resulting stigma, as well as user acceptability to the intervention.

DETAILED DESCRIPTION:
Vesicovaginal fistula (VVF) is a debilitating maternal morbidity that largely results from complications of prolonged, obstructed labor when the trapped fetal head applies direct pressure to pelvic/vaginal tissues and causes widespread ischemia, tissue necrosis, and subsequent extensive fistula formation. Women living with VVF, the most common anatomical presentation of obstetric fistula, experience urinary incontinence which causes discomfort, malodor, and skin infection, as well as social and psychological consequences that increase their vulnerability to the negative effects of stigma and reduce their quality of life.

Traditional management requires surgical repair; however, many women either do not have access to surgery, or access is delayed due to various individual, social, or structural barriers. Non-surgical management, previously explored with non-invasive techniques for residual urinary incontinence, has been under-examined for fistula-related urinary incontinence. The menstrual cup may be a useful option for non-surgical management of obstetric fistula. Clinical and programmatic reports suggest a potential translation of the menstrual cup for collection or control of urine leakage in women with VVF; however, evidence has not been collected and examined systematically within a population in an endemic setting.

While surgical management of fistula remains the gold standard in treatment, research on non-surgical therapies is necessary.Therefore, this study aims to assess the feasibility (including efficacy, safety, and acceptability among users) of using the menstrual cup over a short period among women seeking care for VVF in a clinical setting and, unlike prior reports, includes standardized measures of leakage and prioritizes user perspectives.

A repeated measures design compared volume of leakage with the and without the cup to baseline leakage via a 2-hr pad test among women with VVF seeking surgical repair at a health facility in Ghana. A questionnaire was later administered followed by a physical exam. A paired t-test was used to analyze effect.

Beginning October 2018, semi-structured interviews with up to 24 women seeking treatment at a health facility in Ghana will be carried out on women's experience with fistula, including strategies for coping with urinary incontinence and resulting stigma, as well as their acceptability to the insertable device. This mixed methods approach is necessary to compare quantitative results and qualitative findings regarding what women are already doing to cope with incontinence and stigma, and their acceptability to this device to manage leaking and support coping.

ELIGIBILITY:
Inclusion Criteria:

1. Patient seeking surgical repair for VVF
2. VVF confirmed by gynecologic examination
3. Adequate vaginal capacity to accommodate the menstrual cup
4. Fistula high in vagina (determined at gynecologic examination)
5. Willingness to insert and remove the device by one's self

Exclusion Criteria:

1. Technically difficult to insert and or remove the menstrual cup (eg severely scarred vagina)
2. Unable or unwilling to learn to insert and remove the menstrual cup
3. Patient who declines consent or is incapable of consent
4. Presence of rectovaginal fistula (RVF) or combined RVF and VVF
5. Fistula low in the vagina precluding collection of urine by the menstrual cup

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2019-01-25 (Estimated)

PRIMARY OUTCOMES:
Volume of urinary leakage (in ml) | Over 2 hours
  Measured by 2-hr pad test

SECONDARY OUTCOMES:
Acceptability of the menstrual cup | Over 2 hours
  Using a Likert scale with values ranging from 1-5, acceptability is reported based on ease of use, insertion, wearing, removal, and cleaning. A summarizing acceptability scale is not reported.
Adverse events | Over 2 hours
  Erythema, edema/induration, erosion, bleeding assessed by clinical exam
Rate of enrollment through study completion | through study completion, an average of 1 year
  Number of individuals who enroll out of the total number of individuals screened
Rate of consent through study completion | through study completion, an average of 1 year
  Number of individuals who complete the consent form out of the total number of screened individuals meeting all other inclusion and exclusion criteria
Perceived assessment of leakage with use of the menstrual cup | After 1 hour of use
  Proportion of participants that perceive a reduction in leakage (either marked or slight) with use of the menstrual cup compared to their usual strategy for fistula management. This question uses likert-type responses to note whether the respondent perceives their urine leakage markedly improved, slightly improved, no change, slightly worse, or markedly worse.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel YK Ganyaglo, MPH, MSCI, Principal Investigator — Korle-Bu Teaching Hospital, Accra, Ghana
Locations (1):
- Mercy Women's Catholic Hospital, Mankessim, Central Region, Ghana

IPD SHARING:
Plan to Share IPD: Undecided